CLINICAL TRIAL: NCT01178918
Title: Enhanced Non-Specific T Lymphocytes Response to Influenza A (H1N1) AS03-Adjuvanted Vaccine
Brief Title: Non-specific Response to H1N1 Vaccine
Status: Completed | Type: Observational
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Responsible Party: Principal Investigator, Peter Korošec, Head of Laboratory, The University Clinic of Pulmonary and Allergic Diseases Golnik
Other Study IDs: KOPA-H1N1-01
Record Dates: First submitted 2010-08-04; First posted 2010-08-10 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Influenza H1N1
Keywords: Influenza H1N1; Vaccine; Adjuvant; T Lymphocytes; Non-specific response; Interleukin-2; Non-specific T cell response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers from recipients of H1N1 vaccine

SUMMARY:
This is a prospective observational study with recruitment of healthy volunteers from consecutive recipients of H1N1 influenza vaccine at the University Clinic of Respiratory and Allergic Diseases, Golnik, Slovenia.

The purpose of this study is to evaluate certain safety aspects of adjuvanted influenza H1N1 vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of H1N1 influenza vaccine.
* Healthy individuals with no signs of influenza or other infectious disease.

Exclusion Criteria:

* Signs of influenza or other infectious disease in 1 month before study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers from consecutive recipients of H1N1 influenza vaccine at the University Clinic of Respiratory and Allergic Diseases, Golnik, Slovenia.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12-01 (Actual); Study Completion 2012-07-01 (Actual)

PRIMARY OUTCOMES:
T Cell Immune response monitoring after Influenza A (H1N1) AS03-Adjuvanted Vaccination | At 3 weeks after vaccination
T Cell Immune response monitoring after Influenza A (H1N1) AS03-Adjuvanted Vaccination | At 11 weeks after vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Respiratory and Allergic Diseases, Golnik, Slovenia